CLINICAL TRIAL: NCT04878380
Title: Evaluation of Goal-Based Interventions to Promote and Sustain Healthy Sleep Habits
Brief Title: hiSG Sleep Health Study
Acronym: hiSG-SHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Michael W.L. Chee, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: hiSG-SHS
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Sleep
MeSH Terms: interventions — Organizational Objectives

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tracking (Active Comparator): Throughout the 22 week study, participants in both groups will be rewarded for logging their nightly sleep sessions regularly on their study wearable device, based on a weekly completion bonus for a minimum of 3 nights of sleep preceding weekdays (Sunday - Thursday nights) per week.
  Interventions: Device: Fitbit; Behavioral: Sleep education tips
- Goal-Setting (Experimental): Throughout the 22 week study, participants in both groups will be rewarded for logging their nightly sleep sessions regularly on their study wearable device, based on a weekly completion bonus for a minimum of 3 nights of sleep preceding weekdays (Sunday - Thursday nights) per week.
  During the intervention phase, the Goal-Setting group will be additionally rewarded for achieving sleep goals, i.e. 30 mins longer than their habitual sleep duration and sleeping before midnight.
  Interventions: Device: Fitbit; Behavioral: Sleep education tips; Behavioral: Goal-setting

INTERVENTIONS:
Device: Fitbit — A consumer sleep tracker will be used to monitor sleep patterns throughout the study
Behavioral: Sleep education tips — Sleep tips will be provided before the intervention phase
Behavioral: Goal-setting — During the intervention phase, the Goal-Setting group will be additionally rewarded for achieving sleep goals, i.e. 30 mins longer than their habitual sleep duration and sleeping before midnight.
  Arms: Goal-Setting

SUMMARY:
The hiSG Sleep Health Study seeks to investigate the efficacy of education + goal-based programmes for the promotion of healthy sleep habits and to evaluate its impact on daytime sleepiness and mental health.

DETAILED DESCRIPTION:
This study is a sub-study under the existing Health Insights Singapore study (hiSG). The hiSG study is a longitudinal cohort study among working adults (aged 21-42y), monitoring health parameters through a Fitbit tracker and mobile phone-based questionnaires.

The hiSG Sleep Health Study (hiSG SHS) sub-study, will evaluate the efficacy of two goal-based interventions for improving sleep. Participants will be recruited from the existing hiSG subject pool (target N=300), and should have a habitual sleep duration below the recommended 7h (as determined from the currently available hiSG data). Following informed consent, participants will be randomized by the study team into two groups, a) Goal-Setting and b) Tracking, based on a 2:1 ratio, i.e. in the event 300 participants are enrolled, 200 will be allocated to Goal-Setting and 100 to Tracking.

The study is 22 weeks long and will proceed in 3 main phases, namely, 1) Baseline (Week 1-2) 2) Intervention (Week 3-12), and 3) Follow-up (Week 13-22).

Throughout the study, participants in both groups will be rewarded for logging their nightly sleep sessions regularly on their study wearable device, based on a weekly completion bonus for a minimum of 3 nights of sleep preceding weekdays (Sunday - Thursday nights) per week.

Daily questionnaires probing daytime sleepiness, mood, and stress levels as well as once-per-study phase sleep health, sleep hygiene, work-related stress and mental wellbeing questionnaires will be pushed to participants during the baseline (Week 1-2), intervention (Week 11-12) and follow-up periods (Week 21-22) via the hiSG mobile application. Participants will also be reimbursed for completion of these questionnaires.

Both groups will also receive sleep education tips before the intervention period. During the intervention phase, the Goal-Setting group will be additionally rewarded for achieving sleep goals, i.e. 30 mins longer than their habitual sleep duration and sleeping before midnight.

In addition, given the pervasive telecommuting arrangements presently enforced in many workplaces to curb spread of the COVID-19 pandemic, a work-life balance, burnout and work engagement questionnaire will be administered to better understand reasons that could contribute to poor sleep health and mental wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Existing participants in the hiSG study
* Aged 21-42y
* Sleep <7h habitually on weekdays

Exclusion Criteria:

* Shift workers
* Those required to work in different time zones
* Currently Pregnant
* Nursing mothers

Ages: 21 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration measured by wearable device (mins) | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit longer sleep duration across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in sleep duration regularity (standard deviation) measured by wearable device (mins) | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit more consistent sleep durations across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in bedtimes measured by wearable device | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit earlier bedtimes across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in bedtime regularity (standard deviation) measured by wearable device | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit more consistent bedtimes across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in social jetlag (midpoint of sleep on weekends - weekdays) measured by wearable device | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit reduced social jetlag measures across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in scores on the Sleep Health Index questionnaire | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit improved sleep health across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in scores on the Sleep Hygiene Scale questionnaire | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit better sleep hygiene across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in scores on the Work-Related Perseverative Thought and Work Home Interference questionnaires | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit reduced work stress levels across both Intervention and Follow-Up phases, compared to the Tracking group.
Change in scores on the Oldenberg Burnout Inventory questionnaire | Baseline (Week 1-2), Intervention (Week 11-12), Follow up (Week 21-22)
  We hypothesize that the Goal-Setting group will exhibit reduced burnout across both Intervention and Follow-Up phases, compared to the Tracking group.

SECONDARY OUTCOMES:
Bi-directional relationships between amount of nocturnal sleep obtained and daytime sleepiness levels. | Day-by-day associations (Week 1-2, Week 11-12, Week 21-22)
  We hypothesize that longer sleep duration will be associated with improved next day sleepiness [0-100 scale]
Bi-directional relationships between amount of nocturnal sleep obtained and daytime mood and stress levels. | Day-by-day associations (Week 1-2, Week 11-12, Week 21-22)
  We hypothesize that longer sleep duration will be associated with improved next day stress levels [0-100 scale]
Bi-directional relationships between amount of nocturnal sleep obtained and daytime motivational levels. | Day-by-day associations (Week 1-2, Week 11-12, Week 21-22)
  We hypothesize that longer sleep duration will be associated with improved next day motivational levels [0-100 scale]
Bi-directional relationships between amount of nocturnal sleep obtained and daytime mood levels. | Day-by-day associations (Week 1-2, Week 11-12, Week 21-22)
  We hypothesize that longer sleep duration will be associated with improved next day mood levels [0-100 scale]
Associations between Oldenberg Burnout Inventory, Work-Related Perseverative Thought and Work Home Interference with poorer Sleep Health Index scores. | Average scores (Week 1-2)
  We also hypothesize that individuals who score poorly on these burnout scales will also exhibit poorer sleep health scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Sleep and Cognition, Singapore, Singapore

REFERENCES:
- [Derived] Ong JL, Massar SAA, Lau T, Ng BKL, Chan LF, Koek D, Cheong K, Chee MWL. A randomized-controlled trial of a digital, small incentive-based intervention for working adults with short sleep. Sleep. 2023 May 10;46(5):zsac315. doi: 10.1093/sleep/zsac315. PMID 36546351